CLINICAL TRIAL: NCT04558892
Title: Assessment of Coagulation Disorders and of Enoxaparin's Anti-Xa Activity, When Used for Thromboprophylaxis, in Severe Nephrotic Syndrome.
Brief Title: Anti-Xa Activity of Enoxaparin for Prevention of Venous Thromboembolism in Severe Nephrotic Syndrome.
Acronym: ENOX-inNS
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: The primary objectives were achieved.
Sponsor: Military Institute od Medicine National Research Institute (Other)
Responsible Party: Principal Investigator, Anna Matyjek, Principal Investigator, Military Institute od Medicine National Research Institute
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 5/8952 (443)
Record Dates: First submitted 2020-09-10; First posted 2020-09-22 (Actual); Last update posted 2023-01-30 (Actual); Status verified 2020-09

CONDITIONS: Nephrotic Syndrome
Keywords: Nephrotic syndrome; Enoxaparin; Low molecular weight heparin; Anti-Xa activity; Antifactor Xa; Venous thromboembolism
MeSH Terms: conditions — Nephrotic Syndrome; Venous Thromboembolism | interventions — Enoxaparin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Nephrotic syndrome - fixed dose (NS-FD) (Experimental): Drug: Enoxaparin; Dose: 40 mg; Administration: once daily subcutaneously.
  Interventions: Drug: Enoxaparin
- Nephrotic syndrome - adjusted dose (NS-AD) (Experimental): Drug: Enoxaparin; Dose: 1 mg/kg of ideal body weight; Administration: once daily subcutaneously.
  Interventions: Drug: Enoxaparin
- Control - fixed dose (C-FD) (Active Comparator): Drug: Enoxaparin; Dose: 40 mg; Administration: once daily subcutaneously.
  Interventions: Drug: Enoxaparin

INTERVENTIONS:
Drug: Enoxaparin

SUMMARY:
The primary objective is to test the hypothesis that enoxaparin efficacy is reduced in severe nephrotic syndrome. Another purpose is to compare two dosing regimens.

DETAILED DESCRIPTION:
Nephrotic syndrome (NS) is a rare clinical condition characterized by proteinuria exceeding >3.5 g/24h, hypoalbuminemia, dyslipidemia and edema and is associated with hypercoagulable state. In severe cases, with serum albumin ≤2.5 g/dL, the risk of venous thromboembolic events (VTE) is particularly high, and pharmacological prophylaxis is recommended. However, there is a limited evidence of its efficacy and optimal dosing.

The study is designed as 3 arms clinical trial, with 2 study groups and a single control group. The study groups will include patients with severe NS parallelly, alternately assigned (1:1) into two enoxaparin dosing regimens. The control group will consisted of individuals without proteinuria and edema, similar in terms of age, anthropometric features and renal function to NS patients, who will be administered a standard enoxaparin dose. A peak anti-Xa activity at the steady state will be measured to determine the plasma concentration of enoxaparin. Additional laboratory tests for markers of NS severity, renal function and coagulation system proteins will be performed. The overhydration and body water compartments will be assessed using bioimpedance spectroscopy technique. Nephrotic patients will be followed up by 12 months to assess overt VTE and adverse events associated with enoxaparin use.

ELIGIBILITY:
Inclusion Criteria:

* Severe NS, defined as proteinuria exceeding 3.5 g/24h or 50 mg/kg/24h and serum albumin ≤2.5 g/dL;
* eGFR ≥30 mL/min/1.73 m2.

Exclusion Criteria:

* Body mass index (BMI) ≥40 kg/m2;
* Low body mass (<45 kg for female, <57 kg for male);
* Acute VTE;
* Previously introduced anticoagulation (due to comorbidities);
* Contraindications for enoxaparin;
* Pregnancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2015-10-01 (Actual); Primary Completion 2018-11-30 (Actual); Study Completion 2018-11-30 (Actual)

PRIMARY OUTCOMES:
Therapeutic enoxaparin's anti-Xa activity in nephrotic syndrome. | Average: Day 3-5
  Anti-Xa activity values ≥ 0.3 IU/mL in the steady state of enoxaparin concentration, on average between days 3 and 5.
Minimum threshold of enoxaparin's anti-Xa activity. | Average: Day 3-5
  Anti-Xa activity values ≥ 0.2 IU/mL in the steady state of enoxaparin concentration on average between days 3 and 5.

SECONDARY OUTCOMES:
Severity of nephrotic syndrome. | Day 0, Day 3-5
  Serum or/and urinary concentration of laboratory markers of disease.
Coagulation system protein. | Day 0, Day 3-5
  Plasma concentration or activity of secondary hemostasis system protein (clotting factors, fibrinolysis factors, regulatory molecules).
Renal function. | Day 0, Day 3-5
  Estimated glomerular filtration rate (eGFR) calculated with simplified 4-variable Modification of Diet in Renal Disease (MDRD) formula.
Edema. | Day 0, Day 3-5
  Clinical evaluation of edema using 3-stages scale (I: <5 kg, II: 5-10 kg, III: >10 kg) at enrollment and on the day of measuring anti-Xa activity of enoxaparin.
Overhydration. | Day 3-5
  Overhydration measured by bioimpedance spectroscopy on the day of measuring anti-Xa activity of enoxaparin.

OTHER OUTCOMES:
Venous thromboembolic events. | Follow-up period of 1 year from enrollment.
  Clinically overt episode of VTE.
Adverse events of enoxaparin. | Follow-up period of 1 year from enrollment.
  Episodes of minor and major bleeding or heparin-induced thrombocytopenia.

CONTACTS AND LOCATIONS:
Overall Officials: Anna Matyjek, MD, PhD, Principal Investigator — Military Institute of Medicine
Locations (1):
- Military Institute of Medicine, Warsaw, Masovian District, Poland

REFERENCES:
- [Result] Matyjek A, Rymarz A, Nowicka Z, Literacki S, Rozmyslowicz T, Niemczyk S. Anti-Xa Activity of Enoxaparin for Prevention of Venous Thromboembolism in Severe Nephrotic Syndrome-A Single Center Prospective Study. J Clin Med. 2021 Dec 6;10(23):5709. doi: 10.3390/jcm10235709. PMID 34884411